CLINICAL TRIAL: NCT04577716
Title: The PET-EVAR Study - Predicting Endoleaks Following Endovascular Aortic Aneurysm Repair Using 18F-Sodium Fluoride
Brief Title: Predicting Endoleaks Following Endovascular Aortic Aneurysm Repair Using 18F-Sodium Fluoride
Acronym: PET-EVAR
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other); NHS Lanarkshire (Other Government); NHS Tayside (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC20136
Record Dates: First submitted 2020-09-16; First posted 2020-10-08 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Abdominal Aortic Aneurysm; Endoleak; Stent-Graft Endoleak
Keywords: EVAR; Endoleak; 18F-Sodium Fluoride; PET
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Endoleak | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Aortic tissue specimens obtained from individuals undergoing open surgical repair will be studied histologically, using autoradiography and micro-PET/CT.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Endoleak Group: Participants with a previous Endovascular Aneurysm Repair (EVAR) who have developed an endoleak
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: CT Aortic Angiogram
- No Endoleak Group: Participants with a previous Endovascular Aneurysm Repair (EVAR) who have not developed an endoleak
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: CT Aortic Angiogram
- Pre-EVAR Group: Participants who have an abdominal aortic aneurysm and who are undergoing an Endovascular Aneurysm Repair as standard of care
  Interventions: Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography; Diagnostic Test: 12-month CT Aortic Angiogram; Other: 24-month review

INTERVENTIONS:
Diagnostic Test: 18F Sodium Fluoride Positron Emission Tomography / Computed Tomography — PET scan using the 18F-Sodium Fluoride radiotracer followed by an attenuation correction CT scan
Diagnostic Test: CT Aortic Angiogram — CT scan to assess aortic morphology and contextualise PET scan
  Groups: Endoleak Group; No Endoleak Group
Diagnostic Test: 12-month CT Aortic Angiogram — CT scan to assess aortic morphology and the stent graft
  Groups: Pre-EVAR Group
Other: 24-month review — This will consist of a telephone consultation with the study participant and review of electronic clinical records
  Groups: Pre-EVAR Group

SUMMARY:
The purpose of the study is to describe Sodium Fluoride uptake (using Positron Emission Tomography-Computed Tomography - PET-CT) following Endovascular Aneurysm Repair (EVAR) and to determine whether Sodium Fluoride PET-CT can predict the development of endoleaks.

DETAILED DESCRIPTION:
Abdominal aortic aneurysms are a leading cause of death in the United Kingdom. Surveillance programmes and pre-emptive surgical repair are lifesaving. Traditional open surgical repair is associated with major perioperative morbidity and mortality and there has been a move towards minimally invasive Endovascular Aneurysm Repair (EVAR), which reduces these early risks. However, the cost effectiveness and long-term clinical effectiveness of EVAR is undermined by concerns of durability due to the development of endoleaks and late aneurysm rupture secondary to progression of native aortic aneurysm disease and stent graft failure. It has previously been demonstrated that 18F-Sodium Fluoride Positron Emission Tomography can predict progression of aneurysm disease and is associated with greater rates of abdominal aortic aneurysm expansion and the future risk of rupture or surgical repair.

The investigators here wish to examine whether 18F-Sodium Fluoride on Positron Emission Tomography uptake (i) is increased in patients with endoleaks or related complications, (ii) can prospectively predict the likelihood of developing endoleaks in patients undergoing EVAR, and (ii) is a feasible approach to select patients for EVAR with a reduced future risk of stent graft failure and re-intervention. The investigators believe that there is a compelling scientific rationale for this approach with major translational potential to better select subgroups of patients for EVAR and ultimately improve their outcome.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of AAA as defined by the European Society of Vascular Surgery guidelines on the management of aorto-iliac artery aneurysms, and having undergone endovascular repair within the recommended Instructions For Use (IFU) by the manufacturer. ['Endoleak' and 'No Endoleak groups only]
* Complication will be defined as any type of endoleak or stent graft migration ['Endoleak' group only].
* A diagnosis of AAA requiring endovascular repair OR a diagnosis of juxtarenal AAA requiring fenestrated endovascular aneurysm repair as defined by the European Society of Vascular surgery guidelines on the management of aorto-iliac artery aneurysms and planned EVAR or fenestrated EVAR surgery. ['pre-EVAR' group only]
* Minimum age: 50 years. No maximum age.
* Retain capacity for informed consent

Exclusion Criteria:

* The inability of patients to undergo PET/CT scanning
* Chronic kidney disease (eGFR ≤ 30 mL/min/1.73 m2)
* Major or untreated cancer
* Pregnancy
* Allergy or contra-indication to iodinated contrast
* Inability or unwillingness to give informed consent
* Life-expectancy of less than two years
* Known history of connective tissue disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of individuals with an abdominal aortic aneurysm (AAA). The first part of the study (Study 1 - Case Control Study) will recruit patients with existing EVAR in to two groups: patients that have an endoleak or related complication (endoleak group, n = 22) and those that have remained complication-free (no endoleak group, n = 22). We will also prospectively recruit patients who are yet to receive EVAR or fenestrated EVAR (pre-EVAR group, n = 100) for the (Study 2 - Cohort Study).
  There will be four patient identification centres from which patients will be recruited: NHS Lothian, NHS Lanarkshire, NHS Greater Glasgow and Clyde, and NHS Tayside.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Microcalcification activity in stented and aneurysmal aorta | 12 months
  Will be measured as 18F Sodium Fluoride binding in the aorta. Uptake will be quantified in Standardised Uptake Values and as a tissue to background ratios.

SECONDARY OUTCOMES:
Pattern of microcalcification activity in the stented aorta | 12 months
  Microcalcification activity
Intensity of microcalcification activity in the stented aorta | 12 months
  Microcalcification activity
Endoleaks | 12 months
  Computed tomography and ultrasound endpoints
Stent graft migration | 12 months
  Computed tomography and ultrasound endpoints
Aneurysm sac diameter | 12 months
  Computed tomography and ultrasound endpoints
Neck diameter and neck angulation | 12 months
  Computed tomography and ultrasound endpoints
Geometry: tortuosity, curvature, torsion | 12 months
  Computed tomography and ultrasound endpoints
Aneurysm-related mortality | 24 months
  Clinical endpoints
Re-intervention | 24 months
  Clinical endpoints
All-cause mortality | 24 months
  Clinical endpoints

OTHER OUTCOMES:
Co-localisation of 18F-Sodium Fluoride with histological changes in aortic tissue | 12-36 months
  Uptake of 18F-Sodium Fluoride will be identified on PET-CT scans that are acquired as part of the study visit. This will be compared with histological changes in aortic specimens obtained if participant undergoes an open aortic procedure during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Debono, Principal Investigator — University of Edinburgh
Locations (4):
- United Kingdom (4):
  - Ninewells Hospital, Dundee
  - University Hospital Hairmyres, East Kilbride
  - Royal Infirmary of Edinburgh, Edinburgh
  - Queen Elizabeth University Hospital, Glasgow

IPD SHARING:
Plan to Share IPD: No
There are no plans for individual participant data sharing.

REFERENCES:
- [Result] Debono S, Nash J, Fletcher AJ, Syed M, van Beek EJR, Williams MC, Falah O, Tambyraja A, Dweck MR, Newby DE, Forsythe RO. Aortic sodium [18F]fluoride uptake following endovascular aneurysm repair. Heart. 2023 Oct 26;109(22):1677-1682. doi: 10.1136/heartjnl-2023-322514. PMID 37164479
- [Derived] Debono S, Nash J, Tambyraja AL, Newby DE, Forsythe RO. Endovascular repair for abdominal aortic aneurysms. Heart. 2021 Nov;107(22):1783-1789. doi: 10.1136/heartjnl-2020-318288. Epub 2021 Mar 4. PMID 33674354